CLINICAL TRIAL: NCT00590941
Title: Candidate Gene Polymorphisms and Response to Rituximab-CHOP in Patients With Diffuse Large Cell Lymphoma
Brief Title: Genetic Determinations for Side Effects and Response Rate for Patients Receiving Chemotherapy With Diffuse Large Cell Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 05-0122; 05-0122
Record Dates: First submitted 2007-12-28; First posted 2008-01-11 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Lymphoma; Diffuse Large Cell
Keywords: Lymphoma; Rituximab; CHOP
MeSH Terms: conditions — Lymphoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- R-CHOP (No Intervention): Patients receiving R-CHOP via standard of care which consists of cyclophosphamide 750 mg/m2 IV day 1 of each 21 day cycle, doxorubicin 50 mg/m2 IV day 1 of each 21 day cycle, vincristine 1.4 mg/m2 IV day 1 of each 21 day cycle, prednisone 100 mg PO days 1-5 of each 21 day cycle, and rituximab 375 mg/m2 IV day 1 of each 21 day cycle.
  Interventions: Procedure: Blood draw

INTERVENTIONS:
Procedure: Blood draw — Sample Collection for Genotyping prior to cycle 1 treatment of R-CHOP, if patient is enrolled after cycle 1, sample for genotyping should be collected prior to cycle 2.

SUMMARY:
The purpose of this study is to determine whether people have genes that make them more likely to respond to chemotherapy and/or have side effects from chemotherapy for diffuse large cell lymphoma.

DETAILED DESCRIPTION:
Upon enrollment in the study, patients will have a blood sample collected for genotyping of the FCGR3A gene (immunoglobulin Fc G receptor IIIa), the ABCB1 gene (ATP Binding Cassette Beta 1; also called MDR1), and other candidate genes. Patients will be treated with R-CHOP for six cycles, which is standard therapy for advanced stage DLCL. Response will be monitored by an FDG-PET scan performed after 2 cycles of R-CHOP and restaging exams performed upon completion of chemotherapy. Gene polymorphisms will be analyzed to establish which polymorphisms predict response to R-CHOP.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diffuse large B-cell non-Hodgkin's lymphoma according to the WHO classification, with measurable or evaluable disease
* No prior therapy for NHL. Patient may be enrolled in this study after the first cycle of R-CHOP if all screening evaluations were performed prior to the first cycle of chemotherapy.
* Ann Arbor stage 3 or 4
* Age greater than or equal to 18 years
* Patient must give written informed consent.
* A patient enrolled in another clinical trial may also enroll in this study if the other trial has an R-CHOP treatment arm and the patient is randomized to the R-CHOP only arm. Registration to this study must occur after randomization in the other trial.

Exclusion Criteria:

* CNS involvement
* Known HIV positive
* T-cell lymphoma or history of indolent NHL
* Patients who will be treated with radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2005-02; Primary Completion 2008-07 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Negative [F-18]fluorodeoxyglucose-positron emission tomography (FDG-PET) scan after 2 cycles of R-CHOP | Approximately 42 days (2 cycles of R-CHOP)

SECONDARY OUTCOMES:
Response after six cycles of R-CHOP | Approximately 126 days (6 Cycles of R-CHOP)
Progression free survival | 3 years
Grade 3-4 toxicity | Approximately 156 days

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Cashen, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] A clinical evaluation of the International Lymphoma Study Group classification of non-Hodgkin's lymphoma. The Non-Hodgkin's Lymphoma Classification Project. Blood. 1997 Jun 1;89(11):3909-18. PMID 9166827
- [Background] McKelvey EM, Gottlieb JA, Wilson HE, Haut A, Talley RW, Stephens R, Lane M, Gamble JF, Jones SE, Grozea PN, Gutterman J, Coltman C, Moon TE. Hydroxyldaunomycin (Adriamycin) combination chemotherapy in malignant lymphoma. Cancer. 1976 Oct;38(4):1484-93. doi: 10.1002/1097-0142(197610)38:43.0.co;2-i. PMID 791473
- [Background] Fisher RI, Gaynor ER, Dahlberg S, Oken MM, Grogan TM, Mize EM, Glick JH, Coltman CA Jr, Miller TP. Comparison of a standard regimen (CHOP) with three intensive chemotherapy regimens for advanced non-Hodgkin's lymphoma. N Engl J Med. 1993 Apr 8;328(14):1002-6. doi: 10.1056/NEJM199304083281404. PMID 7680764
- [Background] Vose JM, Link BK, Grossbard ML, Czuczman M, Grillo-Lopez A, Gilman P, Lowe A, Kunkel LA, Fisher RI. Phase II study of rituximab in combination with chop chemotherapy in patients with previously untreated, aggressive non-Hodgkin's lymphoma. J Clin Oncol. 2001 Jan 15;19(2):389-97. doi: 10.1200/JCO.2001.19.2.389. PMID 11208830
- [Background] Coiffier B, Lepage E, Briere J, Herbrecht R, Tilly H, Bouabdallah R, Morel P, Van Den Neste E, Salles G, Gaulard P, Reyes F, Lederlin P, Gisselbrecht C. CHOP chemotherapy plus rituximab compared with CHOP alone in elderly patients with diffuse large-B-cell lymphoma. N Engl J Med. 2002 Jan 24;346(4):235-42. doi: 10.1056/NEJMoa011795. PMID 11807147
- [Background] Habermann TM, Weller EA et al. Phase III Trial of Rituximab-CHOP (R-CHOP) vs. CHOP with a Second Randomization to Maintenance Rituximab (MR) or Observation in Patients 60 Years of Age and Older with Diffuse Large B-Cell Lymphoma (DLBCL). Blood 102: abstract #8, 2003
- [Background] Elstrom R, Guan L, Baker G, Nakhoda K, Vergilio JA, Zhuang H, Pitsilos S, Bagg A, Downs L, Mehrotra A, Kim S, Alavi A, Schuster SJ. Utility of FDG-PET scanning in lymphoma by WHO classification. Blood. 2003 May 15;101(10):3875-6. doi: 10.1182/blood-2002-09-2778. Epub 2003 Jan 16. PMID 12531812
- [Background] Lavely WC, Delbeke D, Greer JP, Morgan DS, Byrne DW, Price RR, Hallahan DE. FDG PET in the follow-up management of patients with newly diagnosed Hodgkin and non-Hodgkin lymphoma after first-line chemotherapy. Int J Radiat Oncol Biol Phys. 2003 Oct 1;57(2):307-15. doi: 10.1016/s0360-3016(03)00599-6. PMID 12957239
- [Background] Zinzani PL, Magagnoli M, Chierichetti F, Zompatori M, Garraffa G, Bendandi M, Gherlinzoni F, Cellini C, Stefoni V, Ferlin G, Tura S. The role of positron emission tomography (PET) in the management of lymphoma patients. Ann Oncol. 1999 Oct;10(10):1181-4. doi: 10.1023/a:1008327127033. PMID 10586334
- [Background] Mikhaeel NG, Timothy AR, O'Doherty MJ, Hain S, Maisey MN. 18-FDG-PET as a prognostic indicator in the treatment of aggressive Non-Hodgkin's Lymphoma-comparison with CT. Leuk Lymphoma. 2000 Nov;39(5-6):543-53. doi: 10.3109/10428190009113384. PMID 11342337
- [Background] Spaepen K, Stroobants S, Dupont P, Vandenberghe P, Thomas J, de Groot T, Balzarini J, De Wolf-Peeters C, Mortelmans L, Verhoef G. Early restaging positron emission tomography with ( 18)F-fluorodeoxyglucose predicts outcome in patients with aggressive non-Hodgkin's lymphoma. Ann Oncol. 2002 Sep;13(9):1356-63. doi: 10.1093/annonc/mdf256. PMID 12196360
- [Background] Jerusalem G, Beguin Y, Fassotte MF, Najjar F, Paulus P, Rigo P, Fillet G. Whole-body positron emission tomography using 18F-fluorodeoxyglucose for posttreatment evaluation in Hodgkin's disease and non-Hodgkin's lymphoma has higher diagnostic and prognostic value than classical computed tomography scan imaging. Blood. 1999 Jul 15;94(2):429-33. PMID 10397709
- [Background] Romer W, Hanauske AR, Ziegler S, Thodtmann R, Weber W, Fuchs C, Enne W, Herz M, Nerl C, Garbrecht M, Schwaiger M. Positron emission tomography in non-Hodgkin's lymphoma: assessment of chemotherapy with fluorodeoxyglucose. Blood. 1998 Jun 15;91(12):4464-71. PMID 9616140
- [Background] Kostakoglu L, Coleman M, Leonard JP, Kuji I, Zoe H, Goldsmith SJ. PET predicts prognosis after 1 cycle of chemotherapy in aggressive lymphoma and Hodgkin's disease. J Nucl Med. 2002 Aug;43(8):1018-27. PMID 12163626
- [Background] Jerusalem G, Beguin Y, Fassotte MF, Najjar F, Paulus P, Rigo P, Fillet G. Persistent tumor 18F-FDG uptake after a few cycles of polychemotherapy is predictive of treatment failure in non-Hodgkin's lymphoma. Haematologica. 2000 Jun;85(6):613-8. PMID 10870118
- [Background] Evans WE, McLeod HL. Pharmacogenomics--drug disposition, drug targets, and side effects. N Engl J Med. 2003 Feb 6;348(6):538-49. doi: 10.1056/NEJMra020526. No abstract available. PMID 12571262
- [Background] Watters JW, McLeod HL. Cancer pharmacogenomics: current and future applications. Biochim Biophys Acta. 2003 Mar 17;1603(2):99-111. doi: 10.1016/s0304-419x(03)00003-9. PMID 12618310
- [Background] McLeod HL, Evans WE. Pharmacogenomics: unlocking the human genome for better drug therapy. Annu Rev Pharmacol Toxicol. 2001;41:101-21. doi: 10.1146/annurev.pharmtox.41.1.101. PMID 11264452
- [Background] Evans WE, Relling MV. Pharmacogenomics: translating functional genomics into rational therapeutics. Science. 1999 Oct 15;286(5439):487-91. doi: 10.1126/science.286.5439.487. PMID 10521338
- [Background] Phillips KA, Veenstra DL, Oren E, Lee JK, Sadee W. Potential role of pharmacogenomics in reducing adverse drug reactions: a systematic review. JAMA. 2001 Nov 14;286(18):2270-9. doi: 10.1001/jama.286.18.2270. PMID 11710893
- [Background] Relling MV, Hancock ML, Rivera GK, Sandlund JT, Ribeiro RC, Krynetski EY, Pui CH, Evans WE. Mercaptopurine therapy intolerance and heterozygosity at the thiopurine S-methyltransferase gene locus. J Natl Cancer Inst. 1999 Dec 1;91(23):2001-8. doi: 10.1093/jnci/91.23.2001. PMID 10580024
- [Background] McLeod HL, Krynetski EY, Relling MV, Evans WE. Genetic polymorphism of thiopurine methyltransferase and its clinical relevance for childhood acute lymphoblastic leukemia. Leukemia. 2000 Apr;14(4):567-72. doi: 10.1038/sj.leu.2401723. PMID 10764140
- [Background] Marsh S, McLeod HL. Thymidylate synthase pharmacogenetics in colorectal cancer. Clin Colorectal Cancer. 2001 Nov;1(3):175-8; discussion 179-81. doi: 10.3816/CCC.2001.n.018. PMID 12450432
- [Background] Ando Y, Saka H, Ando M, Sawa T, Muro K, Ueoka H, Yokoyama A, Saitoh S, Shimokata K, Hasegawa Y. Polymorphisms of UDP-glucuronosyltransferase gene and irinotecan toxicity: a pharmacogenetic analysis. Cancer Res. 2000 Dec 15;60(24):6921-6. PMID 11156391
- [Background] Iyer L, Das S, Janisch L, Wen M, Ramirez J, Karrison T, Fleming GF, Vokes EE, Schilsky RL, Ratain MJ. UGT1A1*28 polymorphism as a determinant of irinotecan disposition and toxicity. Pharmacogenomics J. 2002;2(1):43-7. doi: 10.1038/sj.tpj.6500072. PMID 11990381
- [Background] Park DJ, Stoehlmacher J, Zhang W, Tsao-Wei DD, Groshen S, Lenz HJ. A Xeroderma pigmentosum group D gene polymorphism predicts clinical outcome to platinum-based chemotherapy in patients with advanced colorectal cancer. Cancer Res. 2001 Dec 15;61(24):8654-8. PMID 11751380
- [Background] Alizadeh AA, Eisen MB, Davis RE, Ma C, Lossos IS, Rosenwald A, Boldrick JC, Sabet H, Tran T, Yu X, Powell JI, Yang L, Marti GE, Moore T, Hudson J Jr, Lu L, Lewis DB, Tibshirani R, Sherlock G, Chan WC, Greiner TC, Weisenburger DD, Armitage JO, Warnke R, Levy R, Wilson W, Grever MR, Byrd JC, Botstein D, Brown PO, Staudt LM. Distinct types of diffuse large B-cell lymphoma identified by gene expression profiling. Nature. 2000 Feb 3;403(6769):503-11. doi: 10.1038/35000501. PMID 10676951
- [Background] Rosenwald A, Wright G, Chan WC, Connors JM, Campo E, Fisher RI, Gascoyne RD, Muller-Hermelink HK, Smeland EB, Giltnane JM, Hurt EM, Zhao H, Averett L, Yang L, Wilson WH, Jaffe ES, Simon R, Klausner RD, Powell J, Duffey PL, Longo DL, Greiner TC, Weisenburger DD, Sanger WG, Dave BJ, Lynch JC, Vose J, Armitage JO, Montserrat E, Lopez-Guillermo A, Grogan TM, Miller TP, LeBlanc M, Ott G, Kvaloy S, Delabie J, Holte H, Krajci P, Stokke T, Staudt LM; Lymphoma/Leukemia Molecular Profiling Project. The use of molecular profiling to predict survival after chemotherapy for diffuse large-B-cell lymphoma. N Engl J Med. 2002 Jun 20;346(25):1937-47. doi: 10.1056/NEJMoa012914. PMID 12075054
- [Background] Vitolo U, Botto B, Capello D, Vivenza D, Zagonel V, Gloghini A, Novero D, Parvis G, Calvi R, Ariatti C, Milan I, Bertini M, Boccomini C, Freilone R, Pregno P, Orsucci L, Palestro G, Saglio G, Carbone A, Gallo E, Gaidano G. Point mutations of the BCL-6 gene: clinical and prognostic correlation in B-diffuse large cell lymphoma. Leukemia. 2002 Feb;16(2):268-75. doi: 10.1038/sj.leu.2402349. PMID 11840294
- [Background] Houldsworth J, Olshen AB, Cattoretti G, Donnelly GB, Teruya-Feldstein J, Qin J, Palanisamy N, Shen Y, Dyomina K, Petlakh M, Pan Q, Zelenetz AD, Dalla-Favera R, Chaganti RS. Relationship between REL amplification, REL function, and clinical and biologic features in diffuse large B-cell lymphomas. Blood. 2004 Mar 1;103(5):1862-8. doi: 10.1182/blood-2003-04-1359. Epub 2003 Nov 13. PMID 14615382
- [Background] Hermine O, Haioun C, Lepage E, d'Agay MF, Briere J, Lavignac C, Fillet G, Salles G, Marolleau JP, Diebold J, Reyas F, Gaulard P. Prognostic significance of bcl-2 protein expression in aggressive non-Hodgkin's lymphoma. Groupe d'Etude des Lymphomes de l'Adulte (GELA). Blood. 1996 Jan 1;87(1):265-72. PMID 8547651
- [Background] Cartron G, Dacheux L, Salles G, Solal-Celigny P, Bardos P, Colombat P, Watier H. Therapeutic activity of humanized anti-CD20 monoclonal antibody and polymorphism in IgG Fc receptor FcgammaRIIIa gene. Blood. 2002 Feb 1;99(3):754-8. doi: 10.1182/blood.v99.3.754. PMID 11806974
- [Background] Koene HR, Kleijer M, Algra J, Roos D, von dem Borne AE, de Haas M. Fc gammaRIIIa-158V/F polymorphism influences the binding of IgG by natural killer cell Fc gammaRIIIa, independently of the Fc gammaRIIIa-48L/R/H phenotype. Blood. 1997 Aug 1;90(3):1109-14. PMID 9242542
- [Background] Treon SP, Hansen M, Branagan AR, Verselis S, Emmanouilides C, Kimby E, Frankel SR, Touroutoglou N, Turnbull B, Anderson KC, Maloney DG, Fox EA. Polymorphisms in FcgammaRIIIA (CD16) receptor expression are associated with clinical response to rituximab in Waldenstrom's macroglobulinemia. J Clin Oncol. 2005 Jan 20;23(3):474-81. doi: 10.1200/JCO.2005.06.059. PMID 15659493
- [Background] Maloney DG, Pender-Smith B, et al. Fcg Receptor Polymorphisms Do Not Influence Progression Free Survival of Follicular NHL Patients Treated with CHOP Followed by Rituximab. ASH abstract # 2618, 2004
- [Background] Boettcher S, Pott C, et al. Evidence for Fcg Receptor IIIA-Independent Rituximab Effector Mechanisms in Patients with Follicular Lymphoma Treated with Combined Immuno-Chemotherapy. ASH abstract #2953, 2004
- [Background] Weng WK, Levy R. Two immunoglobulin G fragment C receptor polymorphisms independently predict response to rituximab in patients with follicular lymphoma. J Clin Oncol. 2003 Nov 1;21(21):3940-7. doi: 10.1200/JCO.2003.05.013. Epub 2003 Sep 15. PMID 12975461
- [Background] Dresser MJ. The MDR1 C3435T polymorphism: effects on P-glycoprotein expression/function and clinical significance. AAPS PharmSci. 2001;3(3):4-6. doi: 10.1208/ps0303_commentary3. No abstract available. PMID 11783426
- [Background] Sparreboom A, Danesi R, Ando Y, Chan J, Figg WD. Pharmacogenomics of ABC transporters and its role in cancer chemotherapy. Drug Resist Updat. 2003 Apr;6(2):71-84. doi: 10.1016/s1368-7646(03)00005-0. PMID 12729805
- [Background] Zheng H, Webber S, Zeevi A, Schuetz E, Zhang J, Lamba J, Bowman P, Burckart GJ. The MDR1 polymorphisms at exons 21 and 26 predict steroid weaning in pediatric heart transplant patients. Hum Immunol. 2002 Sep;63(9):765-70. doi: 10.1016/s0198-8859(02)00426-3. PMID 12175731
- [Background] Hoffmeyer S, Burk O, von Richter O, Arnold HP, Brockmoller J, Johne A, Cascorbi I, Gerloff T, Roots I, Eichelbaum M, Brinkmann U. Functional polymorphisms of the human multidrug-resistance gene: multiple sequence variations and correlation of one allele with P-glycoprotein expression and activity in vivo. Proc Natl Acad Sci U S A. 2000 Mar 28;97(7):3473-8. doi: 10.1073/pnas.97.7.3473. PMID 10716719
- [Background] Fellay J, Marzolini C, Meaden ER, Back DJ, Buclin T, Chave JP, Decosterd LA, Furrer H, Opravil M, Pantaleo G, Retelska D, Ruiz L, Schinkel AH, Vernazza P, Eap CB, Telenti A; Swiss HIV Cohort Study. Response to antiretroviral treatment in HIV-1-infected individuals with allelic variants of the multidrug resistance transporter 1: a pharmacogenetics study. Lancet. 2002 Jan 5;359(9300):30-6. doi: 10.1016/S0140-6736(02)07276-8. PMID 11809184
- [Background] Siddiqui A, Kerb R, Weale ME, Brinkmann U, Smith A, Goldstein DB, Wood NW, Sisodiya SM. Association of multidrug resistance in epilepsy with a polymorphism in the drug-transporter gene ABCB1. N Engl J Med. 2003 Apr 10;348(15):1442-8. doi: 10.1056/NEJMoa021986. PMID 12686700
- [Background] Illmer T, Schuler US, Thiede C, Schwarz UI, Kim RB, Gotthard S, Freund D, Schakel U, Ehninger G, Schaich M. MDR1 gene polymorphisms affect therapy outcome in acute myeloid leukemia patients. Cancer Res. 2002 Sep 1;62(17):4955-62. PMID 12208746
- [Background] Juweid ME, Wiseman G, et al. Proc. Am. Soc. of Clin. Onc. 22(14S): 6533, 2004
- [Background] Cheson BD, Horning SJ, Coiffier B, Shipp MA, Fisher RI, Connors JM, Lister TA, Vose J, Grillo-Lopez A, Hagenbeek A, Cabanillas F, Klippensten D, Hiddemann W, Castellino R, Harris NL, Armitage JO, Carter W, Hoppe R, Canellos GP. Report of an international workshop to standardize response criteria for non-Hodgkin's lymphomas. NCI Sponsored International Working Group. J Clin Oncol. 1999 Apr;17(4):1244. doi: 10.1200/JCO.1999.17.4.1244. PMID 10561185
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu